CLINICAL TRIAL: NCT06991504
Title: The Effect of Cervical Stabilization Training and Vestibular Training on Cervical Region and Balance in Individuals With Migraine
Brief Title: The Effect of Cervical Stabilization Training in Individuals With Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, ARZUCAN TOKSAL UÇAR, PhD., Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BEUN-MIGREN
Record Dates: First submitted 2025-05-12; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Migraine
Keywords: migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STABILIZATION GROUP (Experimental): Group receiving cervical stabilization exercise
  Interventions: Behavioral: Cervical Stabilization Exercises
- Vestıbular rehabilitation (Experimental): Group receiving vestibular rehabilitation
  Interventions: Behavioral: vestibular exercises
- Control Group (Experimental): Group receiving classical neck exercise
  Interventions: Behavioral: Classic cervical/ neck exercises

INTERVENTIONS:
Behavioral: Cervical Stabilization Exercises — The main goal of this training is to increase the strength and endurance of the deep cervical flexor and extensor muscles.
  Arms: STABILIZATION GROUP
Behavioral: vestibular exercises — Vestibular exercises are a training used in individuals with migraine to ensure balance and coordination.
  Arms: Vestıbular rehabilitation
Behavioral: Classic cervical/ neck exercises — Classic cervical neck exercises including stretching and strengthening
  Arms: Control Group

SUMMARY:
Studies examining stabilization training and cervical muscle endurance generally focused on headache as the main topic and did not focus on migraine. Studies examining the effects of vestibular training focused on the effects on vestibular migraine and did not address migraine holistically. Although the effects of vestibular rehabilitation and cervical stabilisation training on balance, cervical muscle endurance and joint position error in individuals with migraine have been examined separately, no study has been found in which all these topics were combined. Based on these reasons, this study aims to investigate the effects of two trainings on cervical muscle strength, normal range of motion, anterior tilt, joint position error, deep muscle endurance and balance in individuals with migraine.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being diagnosed with migraine by a neurologist according to the International Headache Society Criteria
* Complaining of headache at least once a week or more in the last year

Exclusion Criteria:

* History of other diseases or operations in the cervical region
* Having any neurological or orthopedic disease
* Passing a serious head and/or neck trauma
* Participating in a physiotherapy program for head and neck pain in the last 12 months
* Having a visual impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-05-03 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Craniovertebral Angle | up to 4 weeks
  Craniovertebral Angle measuremnt
Tragus- Wall Distance | up to 4 weeks
  Tragus- Wall Distance is is used to measure cervical anterior tilt.
Cervical Range of Motion Measurement (C-ROM) | up to 4 weeks
  Cervical Range of Motion Measurement (C-ROM) is used to measure range of motion.
Craniocervical Flexion Test | up to 4 weeks
  Craniocervical Flexion Test measures the endurance of the deep cervical flexor muscles.
Cervical Joint Position Sensation Assessment | up to 4 weeks
  The Cervical Joint Position Sensation Assessment is an easy standardized measurement and provides a sensory assessment.
Mini Balance Assessment Systems Test | up to 4 weeks
  The Mini Balance Assessment Systems Test is an easy-to-administer and reliable balance assessment.

SECONDARY OUTCOMES:
Visual Analogue Scale - VAS | up to 4 weeks
  Visual Analogue Scale - VAS assesses pain.
Pain Catastrophization Scale | up to 4 weeks
  Pain Catastrophization Scale assesses pain.
Migraine-related disability assessment scale | up to 4 weeks
  Migraine-related disability assessment scale is a method applied in migraine patients and evaluates the level of disability.
Neck Disability Questionnaire | up to 4 weeks
  Neck Disability Questionnaire assesses neck disability.
Beck depression questionnaire | up to 4 weeks
  Beck depression questionnaire assesses emotional state

CONTACTS AND LOCATIONS:
Overall Officials: Arzucan Toksal Uçar, PT. PhD:, Principal Investigator — Zonguldak Bulent Ecevit University; Gizem Alarçin, PT., Principal Investigator — Zonguldak Bulent Ecevit University; Esra Acıman Demirel, MD, Principal Investigator — Zonguldak Bulent Ecevit University
Locations (1):
- Zonguldak Bulent Ecevit University, Merkez, Zonguldak Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided